CLINICAL TRIAL: NCT01104948
Title: A Dose Block-randomized, Double-blind, Placebo-controlled, Single/Multiple Dosing, Dose-escalation Clinical Trial to Investigate the Safety, Tolerability, and Pharmacokinetic Characteristics of DA-8031 After Oral Administration in Healthy Male Subjects
Brief Title: A Study to Characterize the Pharmacokinetics of DA-8031 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA-8031
Record Dates: First submitted 2010-04-12; First posted 2010-04-16 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Premature Ejaculatory Dysfunction
MeSH Terms: interventions — DA 8031

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- DA-8031 (Experimental)
  Interventions: Drug: DA-8031
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DA-8031
  Arms: DA-8031
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a dose block-randomized, double-blind, placebo-controlled, single/multiple dosing, dose-escalation study. The study is designed to describe the relationship between multiple doses and pharmacokinetic parameters of DA-8031 as well as safety profile.

ELIGIBILITY:
Inclusion Criteria:

* 20-45 years healthy male subjects
* Body weight :60-90kg, BMI between 18.5-25

Exclusion Criteria:

* show SBP(Systolic Blood Pressure) =<100mmHg or >=140mmHg, or DBP(Diastolic Blood Pressure)=<60mmHg or >=90mmHg, or tachycardia (PR(Pulse Rate)>=100times/min)
* have a history of drug abuse or show positive for drug abuse or cotinine at urine screening
* smokers

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetic parameters such as AUC(Area under concentration-time curve), Cmax, Tmax, T1/2, fe, and CL/F of DA-8031 by as assessment of plasma and urine concentration

SECONDARY OUTCOMES:
To evaluate the safety and tolerance of DA-8031 by assessment of vital signs, clinical laboratory tests, physical examinations, ECG findings, and adverse events collected by investigator questionnaire and subjects spontaneous report

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Institute, Seoul National University Hospital, Seoul, Chongno-Gu, Yon-Gon Dong 28, South Korea